CLINICAL TRIAL: NCT02235558
Title: Super-Selective Intra-Arterial Administration of Verapamil for Neuroprotection After Intra-Arterial Thrombolysis for Acute Ischemic Stroke Phase I Study
Brief Title: Superselective Administration of VErapamil During Recanalization in Acute Ischemic Stroke
Acronym: SAVER-I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Justin Fraser (Other)
Responsible Party: Sponsor-Investigator, Justin Fraser, Asst Professor of Cerebrovascular, Endovascular, and Skull Base Surgery; Departments of Neurological Surgery, Neurology, Radiology, and Anatomy & Neurobiology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0975-F1V
Record Dates: First submitted 2014-09-07; First posted 2014-09-10 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Ischemic Stroke
Keywords: Acute Ischemic Stoke; Thrombectomy; Intraarterial Pharmacotherapy; Neuroprotection
MeSH Terms: conditions — Ischemic Stroke | interventions — Verapamil

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Verapamil (Experimental): Super-selective intra-arterial administration of 10 mg verapamil immediately following successful intra-arterial thrombolysis
  Interventions: Drug: Verapamil

INTERVENTIONS:
Drug: Verapamil — Super-selective intra-arterial administration of 10mg verapamil in 20cc of normal saline will be administered over 20 minutes (1cc/minute) through the microcatheter and into the vessel previously obstructed by clot, immediately following successful intra-arterial thrombolysis. Half-life is 2.8-7.4 hrs.
  Other Names: Isoptin; Verelan; Verelan PM; Calan; Bosoptin; Calaptin; Covera-HS

SUMMARY:
The purpose of this study is to determine whether super-selective intra-arterial administration of verapamil immediately following successful intra-arterial thrombolysis is safe as a potential neuroprotective agent. Standard procedures are cerebral angiography and intra-arterial thrombolysis (intra-arterial administration of tPA and/or mechanical thrombectomy). Experimental procedure is superselective injection of verapamil intra-arterially.

DETAILED DESCRIPTION:
This trial represents the first time that verapamil will be evaluated in human subjects as a superselectively administered neuroprotective agent administered in an acute time frame as an adjunct to intra-arterial thrombolysis. The methods for administration, along with the routinized followup, will provide a paradigm for studying other potential neuroprotective agents. Subjects will undergo cerebral angiography with intra-arterial thrombolysis, which is standard of care. 'Intra-arterial thrombolysis will include possible intra-arterial administration of tPA, as well as possible mechanical thrombectomy with an accepted thrombectomy device. This includes the Mercí Retriever (Concentric Medical, Mountain View, CA), the Penumbra System (Penumbra, Alameda, CA), the Solitaire stent-triever (EV3, Covidien, Irvine, CA), and the Trevo stent-triever (Concentric Medical, Mountain View, CA). Immediately after the intra-arterial thrombolysis component of the angiographic procedure is completed, the microcatheter used during the procedure will be left in or guided into the vessel location of the clot. 10mg of verapamil in 20cc of normal saline will be administered over 20 minutes (1cc/minute) through the microcatheter and into the vessel previously obstructed by clot. At the conclusion of infusion, the microcatheter will be removed. Angiography through the guide catheter of the cerebral circulation in question will be performed to ensure no new thromboembolic event from the microcatheterization (standard of care). The catheters will be removed, and the arterial puncture site closed in the standard fashion. Patients will receive a noncontrast CT scan or MRI approximately 24 hours after intervention to determine the presence or absence of intracerebral hemorrhage (ICH) after intervention. This would be considered standard practice for intra-arterial thrombolysis. Both imaging studies can detect ICH, and the choice of one or the other will be determined by clinical criteria; CT or MRI may be preferable for different reasons depending upon the patient's clinical scenario. The determination of hemorrhage will be made by the official dictation of a diagnostic neuroradiologist not directly involved in the study. The hemorrhage will be considered an adverse event if it is deemed symptomatic in accordance with the criteria used in the International Management of Stroke (IMS) III study. Briefly, a hemorrhage is defined as symptomatic if occurring within 24+/-6 hours after study inclusion, temporally related to the intervention, and occurs with worsening neurological status as documented in the clinical exam. A 4 point or more increase in the NIHSS stroke scale would qualify as a significant worsening in status. Furthermore, hemorrhage that requires intervention surgically or endovascularly would be deemed significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 21-85 years old, male or female
2. Suspected acute ischemic stroke based on clinical and radiographic evidence as determined and documented by the Stroke Neurology team at University of Kentucky.
3. Patients must meet criteria for intra-arterial thrombolysis as determined and documented by Interventional Neuroradiology attending physician (JF or AA).
4. Patients must have an acute thromboembolus within an intracranial artery (internal carotid, anterior cerebral, middle cerebral, posterior cerebral, basilar, vertebral) which undergoes pharmacologic (tissue plasminogen activator - tPA) and/or mechanical (eg. Merci or Penumbra clot retrieval) thrombolysis.
5. Patients with impaired capacity may be included, as the pathology to be studied (stroke) may impair their capacity (please see attached required documentation regarding impaired capacity).
6. Patients must have a TICI 2A or better revascularization via intra-arterial thrombolysis.

For reference, the TICI Scale is defined below:

0 = No Perfusion

1. = Perfusion past the initial obstruction but limited distal branch filling with little or slow distal perfusion
2. A = Perfusion of less than 50% of the vascular distribution of the occluded artery

2B = Perfusion of 50% or greater (but not complete) of the vascular distribution of the occluded artery 3 = Full perfusion with filling of all distal branches

Exclusion Criteria:

1. Pregnant women (would not qualify for intra-arterial thrombolysis as standard of care).
2. Patients who undergo intra-arterial thrombolysis for acute stroke, in whom only TICI 0 or 1 revascularization is obtained.
3. Patients with occlusion of the cervical common or internal carotid artery will be excluded from the study.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the presence or absence of intracranial hemorrhage | 24-48 hours after treatment
  Patients will receive a noncontrast CT scan or MRI approximately 24 hours after intervention to determine the presence or absence of intracerebral hemorrhage (ICH) after intervention.

SECONDARY OUTCOMES:
Absence of intracranial hemorrhage | At follow-up intervals: Day 30 ± 14 days, 3 Months ± 30 days, 6 Months ± 30 days, 12 Months± 30 days
  Improved clinical outcomes at followup intervals as measured by the modified Rankin score.

OTHER OUTCOMES:
Absence of systemic side effects of verapamil administration | 24-48 hours
  Patients will receive a noncontrast CT scan or MRI approximately 24 hours after intervention to determine the presence or absence of intracerebral hemorrhage (ICH) after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Justin F. Fraser, MD, Principal Investigator — University of Kentucky Department of Neurological Surgery
Locations (1):
- University of Kentucky Deparment of Neurosurgery, UK Chandler Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No